CLINICAL TRIAL: NCT03290456
Title: A Prospective, Multicentric, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Remission MAINtenance Using Extended Administration of Prednisone in Systemic Anti-neutrophil Cytoplasmic Antibodies (ANCA)-Associated Vasculitis.
Brief Title: Evaluate the Remission MAINtenance Using Extended Administration of Prednisone in Systemic Anti-neutrophil Cytoplasmic Antibodies (ANCA)-Associated Vasculitis.
Acronym: MAINEPSAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 69HCL17_0020
Record Dates: First submitted 2017-08-24; First posted 2017-09-25 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Granulomatosis With Polyangitis
Keywords: Vasculitis; GPA; Granulomatosis with Polyangitis; MPA; Microscopic Polyangitis; Systemic anti-neutrophil cytoplasmic antibodies (ANCA); Prednisone; glucocorticoids; Remission Maintenance; Rituximab; Cyclophosphamide
MeSH Terms: conditions — Vasculitis | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prednisone 5mg/day extended of 12 additional months (Experimental): Prednisone 5mg/day will be administered from Day 1 to Month 12
  Interventions: Drug: Prednisone 5mg/day extended of 12 additional months
- Placebo 5mg/day extended of 12 additional months (Placebo Comparator): Placebo 5mg/day will be administered from Day 1 to Month 12
  Interventions: Drug: Placebo 5mg/day extended of 12 additionnal months.

INTERVENTIONS:
Drug: Prednisone 5mg/day extended of 12 additional months — Prednisone 5mg/day orally during 12 Month + 1 mg/week tapering until 0mg.
  Arms: Prednisone 5mg/day extended of 12 additional months
Drug: Placebo 5mg/day extended of 12 additionnal months. — 1mg/week orally tapering Prednisone until Month 1 + Placebo orally 5mg/day until Month 13
  Arms: Placebo 5mg/day extended of 12 additional months

SUMMARY:
Immunosuppressive therapy of granulomatosis with polyangiitis (GPA, Wegener's) and microscopic polyangiitis (MPA) has transformed the outcome from death to a strong likelihood of disease control and temporary remission. However, most patients have recurrent relapses that lead to damage and require repeated treatment associated with long-term morbidity and death.

Rituximab has been shown to be as effective as cyclophosphamide to induce remission and maintenance of remission in severe GPA and MPA patients, with an acceptable safety profile . Although rituximab is becoming the standard of care for maintenance therapy in these patients, relapse still occurs and the optimal duration of prednisone therapy remains debated.

On the one hand, most US studies use early withdrawal (6-12 months) because of feared side effects. On the other hand, most European trials propose late withdrawal (>18 months) given a lower observed relapse rate on long-term low dose glucocorticoids treatment.

In a systematic review and meta-analysis, glucocorticoids regimen was the most significant variable explaining the variability between the proportions of ANCA-associated vasculitis patients with relapses. Nevertheless, it was an indirect estimation of treatment effect because of the absence of dedicated randomized trial. This meta-analysis concluded that combined longer-term (i.e. >12 months) use of low dose prednisone or nonzero glucocorticoids target is associated with a 20% reduction of relapse compared to early withdrawal (i.e. ≤12 months).

The relapse rate in patients with early glucocorticoids (10-12 months) withdrawal was provided in two studies and was of 37 and 34%, respectively. By contrast, the relapse rate in patients with late prednisone withdrawal (18-24 months) and receiving rituximab as maintenance treatment was 14% at 24 months in the MAINRITSAN trial. Of note, the decision to withdraw glucocorticoids after 18 months was left to physician's discretion in this study and two thirds of the nonsevere relapses occurred when patients were off prednisone.

The trial detailed here is the first prospective trial evaluating the length of glucocorticoid administration as remission adjunctive treatment for patients with GPA or MPA.

DETAILED DESCRIPTION:
Immunosuppressive therapy of granulomatosis with polyangiitis (GPA, Wegener's) and microscopic polyangiitis (MPA) has transformed the outcome from death to a strong likelihood of disease control and temporary remission. However, most patients have recurrent relapses that lead to damage and require repeated treatment associated with long-term morbidity and death.

Rituximab has been shown to be as effective as cyclophosphamide to induce remission and maintenance of remission in severe GPA and MPA patients, with an acceptable safety profile. Although rituximab is becoming the standard of care for maintenance therapy in these patients, relapse still occurs and the optimal duration of prednisone therapy remains debated.

On the one hand, most US studies use early withdrawal (6-12 months) because of feared side effects. On the other hand, most European trials propose late withdrawal (>18 months) given a lower observed relapse rate on long-term low dose glucocorticoids treatment.

In a systematic review and meta-analysis, glucocorticoids regimen was the most significant variable explaining the variability between the proportions of ANCA-associated vasculitis patients with relapses. Nevertheless, it was an indirect estimation of treatment effect because of the absence of dedicated randomized trial. This meta-analysis concluded that combined longer-term (i.e. >12 months) use of low dose prednisone or nonzero glucocorticoids target is associated with a 20% reduction of relapse compared to early withdrawal (i.e. ≤12 months).

The relapse rate in patients with early glucocorticoids (10-12 months) withdrawal was provided in two studies and was of 37 and 34%, respectively. By contrast, the relapse rate in patients with late prednisone withdrawal (18-24 months) and receiving rituximab as maintenance treatment was 14% at 24 months in the MAINRITSAN trial. Of note, the decision to withdraw glucocorticoids after 18 months was left to physician's discretion in this study and two thirds of the nonsevere relapses occurred when patients were off prednisone.

The trial detailed here is the first prospective trial evaluating the length of glucocorticoid administration as remission adjunctive treatment for patients with GPA or MPA.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of MPA or GPA independently of ANCA status,
* Patient aged of 18 years or older,
* Patients with newly-diagnosed disease or relapsing disease at the time of screening, with an inactive disease defined as a BVAS = 0,
* Patients receiving maintenance infusion of rituximab 500 mg at 6 and 12 months after the start of vasculitis induction
* Patients receiving 5-10 mg/day of prednisone at screening,
* Patient able to give written informed consent prior to participation in the study.
* At Inclusion visit day, patient must be between 5 and 10 mg/day prednisone and at randomization visit day (D1), patient must be at 5 mg/day prednisone

Exclusion Criteria:

* Patients with EGPA, or other vasculitides, defined by the ACR criteria and/or the Chapel Hill Consensus Conference,
* Patients with vasculitis with active disease defined as a BVAS >0,
* Patients with acute infections or chronic active infections (including HIV, HBV or HCV),
* Patients with active cancer or recent cancer (<5 years), except basocellular carcinoma and prostatic cancer of low activity controlled by hormonal treatment,
* Pregnant women and lactation. Patients with childbearing potential should have reliable contraception for the all duration of the study,
* Patients with other uncontrolled diseases, including drug or alcohol abuse, severe psychiatric diseases, that could interfere with participation in the trial according to the protocol,
* Patients included in other investigational therapeutic study within the previous 3 months,
* Patients suspected not to be observant to the proposed treatments,
* Patients who have white blood cell count ≤4,000/mm3,
* Patients who have platelet count ≤100,000/mm3,
* Patients who have ALT or AST level greater than 3 times the upper limit of normal that cannot be attributed to underlying MPA-GPA disease,
* Patients unable to give written informed consent prior to participation in the study.
* Patients with contraindication to use rituximab,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2029-10-20 (Estimated); Study Completion 2029-10-20 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival, relapse being defined as BVAS > 0. | from Screening to Month 30.
  rate of relapse-free survival of patients continuing low-dose prednisone treatment until Month 10 VS those who will have prednisone treatment cessation at Month 1, on remission maintenance with Rituximab therapy, after achievement of remission of GPA or MPA, defined as a survival of patients maintaining a BVAS=0 at Month 30, in patient with newly-diagnosed or relapsing GPA or MPA and who will all have received glucocorticoids for 12 months after diagnosis or last flare before inclusion.

SECONDARY OUTCOMES:
Compare the rate of serious adverse events between Inclusion and Month 30 after randomization | from Day 1 to Month 30
  Proportion of patients with at least one adverse event between inclusion and Month 30.
  * Percentage of patients with at least one serious adverse event between inclusion and Month 30, corresponding to any adverse event that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity or congenital anomaly/birth defect or any other adverse event considered "medically significant".
  * Number of deaths, whatever the cause at Month 30.
Compare the rate of predefined severe events related to glucocorticoids between inclusion and Month 30 including osteoporotic fracture and weight gain. | From Screening to Month 30
  Percentage of patients with at least one predefined severe event corresponding to adverse events of grade 3 to 5 of the Common Terminology Criteria, including severe side effect related to glucocorticoids (infection requiring hospitalization or intravenous antibiotics, osteoporotic fracture, diabetes requiring medication, cardiovascular event, symptomatic osteonecrosis, psychiatric or mood disorder requiring drug administration, weight gain >10 kg) between inclusion and Month 30
  - Weight gain between inclusion and Month 30
To compare the rate of vasculitis relapse at Month 30 | from Day 1 to Month 30
  Proportion of patients with minor or major vasculitis relapse between inclusion and Month 30 (BVAS >0) and time to first vasculitis relapse
To compare the prednisone use between inclusion and Month 30 | from screening to Month 30
  Prednisone area under the curve of administrated dose between inclusion and Month 30
To compare variation of the Bone mineral density and markers between inclusion and Month 30 | From Screening to Month 30
  Variation of the Bone mineral density between inclusion and Month 30
  - Variation of the Bone markers including C-terminal crosslinked telopeptide of type I collagen (CTX) and serum procollagen type 1 amino-terminal propeptide (P1NP) between inclusion and Month 30
To compare sequelae assessed by BVAS (vasculitis activity) at 30 months | From Screening to Month 30.
  BVAS (vasculitis activity) at 30 months
  - Variation of BVAS (Vasculitis activity)
To compare sequelae assessed by the Vasculitis Damage Index (VDI) at 30 months | From screening to Month 30.
  * Vasculitis Damage Index at 30 months
  * Variation of VDI,
- To compare sequelae assessed by Combined Damage Assessment Index (CDA) at 30 months | From Screening to Month 30.
  * Combined Damage Assessment Index at 30 months
  * Variation of CDA (damage),
- To compare functional disability at Month 30 after randomization (Day 1) in both arms | From Day 1 to Month 30.
  Variation of HAQ (disability) between inclusion and at Month 30
To compare quality of life at Month 30 after randomization (Day 1) in both arms | - From Day 1 to Month 30.
  - Variation of SF-36 (quality of life) between inclusion and at Month 30
- To compare healthcare resource utilization at Month 30 after randomization (Day 1) in both arms | From Day 1 to Month 30.
  - Healthcare resource utilization between inclusion and Month 30 being defined as the percentage of patients being hospitalized at least once except only for rituximab infusions

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe LEGA, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (41):
- France (41):
  - CHU Amiens-Hôpital Nord, Amiens
  - CHU Angers, Angers
  - Clinique Rhône-Durance, Avignon
  - Hôpital Jeanne d'Arc, Bar-le-Duc
  - Hôpital Avicenne, Bobigny
  - Hôpital La Cavale Blanche, Brest
  - Hôpital Louis Pradel, Bron
  - CHU de Caen - Cote de Nacre, Caen
  - Hôpital Louis Pasteur, Chartres
  - CHU Estaing, Clermont-Ferrand
  - CHU Gabriel Montpied, Clermont-Ferrand
  - CHIC Créteil, Créteil
  - CHRU François Mitterrand, Dijon
  - CHRU Lille - Hôpital Claude Huriez, Lille
  - Centre Hospitalier Croix Rousse, Lyon
  - Hôpital Edouard Herriot, Lyon
  - Hôpital de la Conception, Marseille
  - Hôpital La Timone, Marseille
  - HP Site Belle Isle, Metz
  - CHU Nantes - Hôtel Dieu, Nantes
  - CHU de Nice - Hôpital Pasteur 2, Nice
  - Hôpital la Pitié Salpêtrière, Paris
  - Hôpital Cochin, Paris
  - Hôpital Européen G. Pompidou, Paris
  - Hôpital Saint Louis, Paris
  - Hôpital Haut Lévêque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CH Lyon Sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - CHRU Rennes - Hôpital Sud, Rennes
  - Hôpital Charles Nicolle, Rouen
  - CHU Strasbourg, Strasbourg
  - CHRU Hautepierre, Strasbourg
  - Hopitaux Universaitaire de Strasbourg Hopitaux, Strasbourg
  - Hôpital Foch, Suresnes
  - CHRU Bretonneau, Tours
  - CH de Troyes, Troyes
  - CH Valenciennes, Valenciennes
  - Hôpitaux de Brabois, Vandœuvre-lès-Nancy
  - CH Bretagne Atlantique, Vannes
  - CH de Verdun, Verdun

IPD SHARING:
Plan to Share IPD: No